CLINICAL TRIAL: NCT06696534
Title: Exploring Participant Preference for Screening Methods and Experience Into Colorectal Cancer Screening Programme
Acronym: MS-Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ADVANCED MARKER DISCOVERY S.L. (Industry)
Collaborators: SERMAS (Unknown); ULS de Santa Maria (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AMD-CCR-2024-01; 2024-NDMH-5101_240046 (Other Grant/Funding Number: EIT-Health)
Record Dates: First submitted 2024-11-12; First posted 2024-11-20 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Screening for Colon Cancer; Survey and Questionnaire
Keywords: colorectal cancer; screening programme; experience; preference; questionnaire
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FIT/FOBT population (Other): Average-risk population undergoing FIT/FOBT within the colorectal cancer screening programme.
  Interventions: Other: Survey using a questionnaire.

INTERVENTIONS:
Other: Survey using a questionnaire. — Preference questionnaire for colorectal cancer screening methods
Other: Survey using a questionnaire. — Experience questionnaire into colorectal cancer screening programme

SUMMARY:
The goal of this low-risk interventional study is to analyze participants' assessment of colorectal cancer screening program through screening method preference and experience after FOBT analysis in screaned participant population for colorectal cancer; could include any of the following: both sexes, age 50-69 years, asympthomatic volunteers. The main aims to answer are:

* Values of experience of participants into screening programme.
* Values of preferences of participants for screening methods.

Participants will answer two questionnaires and they'll be given their information and clinical data to investigator or health personnel.

ELIGIBILITY:
Inclusion Criteria:

* Participants ages from 50 to 69 years (both included) at the time of informed consent signed.
* Participants invited to participate in population-based screening programme who are eligible to undertake FOBT at the Primary Health Care Center.
* Participants should sign an informed consent. They must understand the nature, significance, implications, and risks of the clinical study before signing the informed consent form.

Exclusion Criteria:

* Participants who have not delivery a stool sample in the Primary Health Care Center before signing the informed consent form.
* Participants with a previous colonoscopy in consequence of a FOBT positive result.
* Participants who are in a dependent personal or non-medical relationship with the Sponsor or the Investigators.

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Value of questionnaires into screening programme | 12 months
  The percentage of number of answers from each experience and preference questions

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Perez, MD, Principal Investigator — Primary Health Care Centre Mar Báltico; Ana Rita, MD, Principal Investigator — Unidade Local de Saúde de Santa Maria
Locations (2):
- UCSP Sete Rios, Lisbon, Portugal
- CS Mar Báltico, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adler A, Geiger S, Keil A, Bias H, Schatz P, deVos T, Dhein J, Zimmermann M, Tauber R, Wiedenmann B. Improving compliance to colorectal cancer screening using blood and stool based tests in patients refusing screening colonoscopy in Germany. BMC Gastroenterol. 2014 Oct 17;14:183. doi: 10.1186/1471-230X-14-183. PMID 25326034
- [Background] De Angelis R, Demuru E, Baili P, Troussard X, Katalinic A, Chirlaque Lopez MD, Innos K, Santaquilani M, Blum M, Ventura L, Paapsi K, Galasso R, Guevara M, Randi G, Bettio M, Botta L, Guzzinati S, Dal Maso L, Rossi S; EUROCARE-6 Working Group. Complete cancer prevalence in Europe in 2020 by disease duration and country (EUROCARE-6): a population-based study. Lancet Oncol. 2024 Mar;25(3):293-307. doi: 10.1016/S1470-2045(23)00646-0. Epub 2024 Jan 30. PMID 38307102
- [Background] Siegel RL, Wagle NS, Cercek A, Smith RA, Jemal A. Colorectal cancer statistics, 2023. CA Cancer J Clin. 2023 May-Jun;73(3):233-254. doi: 10.3322/caac.21772. Epub 2023 Mar 1. PMID 36856579